CLINICAL TRIAL: NCT07130045
Title: Effect of Hybrid Endurance and Strength Training (HyBEST) on Health-Related Outcomes and Quality of Life in Patients With Coronary Artery Disease During Phase II Cardiac Rehabilitation Program
Brief Title: Hybrid Exercise Program for Heart Disease: Effect on Health and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025116-14608; FRGS/1/2023/SS10/UITM/03/4 (Other Grant/Funding Number: MALAYSIAN FUNDAMENTAL RESEARCH GRANT SCHEME)
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
Keywords: coronary artery disease; combined training; hybrid; cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Endurance and Strength Training (HybEST) (Experimental): HybEST will be delivered three times weekly over eight weeks; there will be two supervised sessions at the center and 22 unsupervised sessions at home.
  Interventions: Other: Hybrid Endurance Strength Training
- Usual Care (UC) (Active Comparator): The UC group participants will participate in combined endurance and strength training similar to the intervention group's weekly center-based session over eight weeks.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Hybrid Endurance Strength Training — HybEST will be delivered three times weekly over eight weeks, with two supervised sessions at the center and 22 unsupervised sessions at home. The exercise characteristics of supervised HybEST and unsupervised HybEST are described. Monitoring methods for unsupervised HybEST include a wearable tracking device that collects data on patients' health parameters (arterial oxygen saturation (SpO2), heart rate, and blood pressure) and weekly phone calls. The unsupervised sessions will include video material on the home-based exercise program.
  Other Names: HyBEST
  Arms: Hybrid Endurance and Strength Training (HybEST)
Other: Usual Care — The UC group participants will participate in combined endurance and strength training similar to the intervention group's weekly center-based session over eight weeks.
  Other Names: UC
  Arms: Usual Care (UC)

SUMMARY:
Cardiac rehabilitation (CR) participation remains suboptimal, partly due to logistical challenges and limited access to center-based programs. Hybrid Endurance-Strength Training (HybEST) offers an alternative model by combining supervised endurance and strength exercises with home-based components. The main questions it aims to answer are:

* Does a hybrid exercise program significantly improve a patient's body function and structures [exercise capacity, body composition, and muscle strength] compared to usual care?
* Does a hybrid exercise program significantly improve a patient's activity [functional capacity, physical activity, and total energy expenditure] compared to usual care?
* Does a hybrid exercise program significantly improve a patient's participation [health-related quality of life] compared to usual care?

This single-center, two-arm parallel randomized clinical trial aims to evaluate the effects of HybEST on health-related outcomes and quality of life among patients with coronary artery disease in Phase II CR. Eligible participants will be randomly assigned in a 1:1 ratio to either the HybEST intervention group or the standard CR control group using a lottery method, specifically the sealed envelope approach. Assessments will be conducted at baseline (T0), Week 5 (T2), and Week 9 (T3) to measure changes in health-related outcomes and quality of life.

DETAILED DESCRIPTION:
In recent years, models for delivering cardiac rehabilitation (CR) have advanced by incorporating structured exercise methods and technology into routine practice. Hybrid Endurance-Strength Training (HybEST) combines supervised center-based sessions with home-based elements, supported by digital tools such as remote monitoring and virtual consultations. This hybrid approach may help overcome common barriers to CR participation, including travel distance, scheduling conflicts, and work commitments. This single-centre, two-arm parallel randomized controlled trial aims to evaluate the effects of a hybrid exercise program in patients with coronary heart disease. The objectives are;

* To evaluate the effects of a hybrid exercise program on patients' body function and structures, including exercise capacity, body composition, and muscle strength, compared to usual care.
* To determine the effects of a hybrid exercise program on patients' activity, including functional capacity, physical activity, and total energy expenditure, compared to usual care.
* To assess the effects of a hybrid exercise program on patients' participation, specifically health-related quality of life, compared to usual care.

A total of 84 eligible participants (42 per group, accounting for 14% attrition) will be randomized into either the intervention or control group. The usual care group will follow a standard exercise program consisting of endurance and strength components. This program includes supervised exercise sessions at the center once a week for eight weeks, along with educational materials on exercising at home. The intervention group will participate in a hybrid training program that combines endurance and strength training over eight weeks. Their program includes two supervised sessions at the center and 22 unsupervised sessions at home. Participants will receive exercise educational videos via WhatsApp (Weeks 1-8) and a fitness tracker to support unsupervised sessions. Weekly virtual follow-ups will be conducted from Week 1 to Week 8. Outcome measures include Exercise Capacity, Body Composition, Muscle Strength, Physical Activity and METs, Barrier Scales, and Health-Related Quality of Life. Data will be analyzed using IBM SPSS version 26.0, with statistical significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older.
* Diagnosed with coronary artery disease (CAD), with or without invasive treatment, maintaining a normal sinus rhythm and preserved left ventricular ejection fraction (LVEF).
* In a stable clinical condition.
* capable of regularly attending a supervised exercise program.
* Able to complete questionnaires in English or Malay.

Exclusion Criteria:

* They exhibited abnormal responses during the initial exercise test, such as irregular haemodynamic responses, ST segment depression greater than 2 mm, or any ventricular fibrillation.
* Their forced expiratory volume in 1 second (FEV1) or forced vital capacity (FVC) is less than 50% of the predicted value.
* They cannot participate in exercise testing due to non-cardiac limitations.
* They have been hospitalized due to heart failure within the past year.
* They have uncontrollable hypertension.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Treadmill stress test | Day 0, Week 9
  A treadmill stress test will be used to assess the participant's exercise capacity. This type of stress testing is typically performed with the Bruce protocol on either a treadmill or an ergometer, monitored with electrocardiography (ECG) and blood pressure. The Bruce protocol requires participants to complete successive 3-minute stages, with each stage increasing in walking speed and incline. During the test, data on heart rate (HR), blood pressure (BP), and ECG changes will be recorded at the end of each stage. After testing, a report will be generated outlining (i) ECG interpretation and baseline HR and BP, (ii) exercise-induced changes in ECG, (iii) maximum heart rate and blood pressure during exercise, (iv) estimated exercise capacity in metabolic equivalents (METs), (v) exercise duration and stage completed, and (vi) symptoms experienced during exercise and reasons for test termination.

SECONDARY OUTCOMES:
Body composition | Day 0, Week 5, Week 9
  Body composition, including body mass index (BMI), body fat percentage, lean mass percentage, and weight in kilograms, will be measured using the bioimpedance meter (OMRON HBF-500INT). Participants' height (meters) will be recorded with the SECA stadiometer. To determine waist circumference, the midpoint between the front-back hip bone and the bottom rib border will be identified when the subject is upright. The average will be calculated by dividing the sum of the two measurements by two.
Muscle strength | Day 0, Week 5, Week 9
  The strength of major muscles in the upper and lower limbs will be measured using a handheld dynamometer (HHD). A plinth-mounted seat and armrest are provided for the participant's positioning and restraint during HHD testing.
Functional Capacity | Day 0, Week 5, Week 9
  The goal of the Six-Minute Walk Test (6MWT) is for participants to walk as far as they can at a comfortable pace. Every minute, patients will receive standardized encouragement such as "You are doing well" or "Keep up the good work," along with a reminder of the remaining time. Qualified personnel will walk behind the patient to supervise the test. During the test, patients are allowed to stop if necessary, but they will be advised to resume walking as soon as possible. Patients may use their walking aids during the test, and 6MWD will be recorded in meters. Heart rate (HR) and oxygen saturation (SpO2) will be measured before, during, and after the 6MWT using pulse oximetry (Model 2500, Nonin Medical, Inc., Minneapolis, MN, USA).
Physical Activity | Day 0, Week 5, Week 9
  The International Physical Activity Questionnaire (IPAQ) will be used to assess the level of physical activity based on information about the time spent walking, participating in moderate-to-vigorous activities, and avoiding sedentary behavior during the previous seven days. According to participant responses, physical activity is categorized into three levels: moderate (600-3000 MET minutes/week), vigorous (more than 3000 MET minutes/week), and light (less than 600 MET minutes/week).
Total Energy Expenditure | Day 0, Week 5, Week 9
  METs will be assessed using a treadmill stress test conducted according to standard protocols (e.g., Bruce or Modified Bruce). Participants will exercise until they reach volitional fatigue or achieve predetermined termination criteria based on clinical guidelines. The highest workload achieved, expressed in METs, will be calculated from the treadmill speed and grade at peak exercise.
Health-related Quality of Life | Day 0, Week 9
  The Medical Outcomes Study Short Form Health Survey (SF-36) will be used to evaluate a person's health status. The SF-36 questionnaire is a standardized tool with 36 items that measure eight different subscales, which cover various aspects of physical functioning, role functioning, physiological discomfort, general health, vitality, social functioning, role-emotional, and mental health. Both individual subscale scores and two summary scores, known as the physical component summary score (PCS) and mental component summary score (MCS), can be calculated.
Self-efficacy | Day 0, Week 9
  The Self-efficacy to Exercise (SEE) questionnaire consists of nine items. The overall score is the sum of all answers to these questions, with total scores ranging from 0 to 90. A higher score indicates greater self-efficacy for exercising.
Barriers to participation | Day 0, Week 9
  To identify barriers to CR participation, participants will complete a self-administered Cardiac Rehabilitation Barriers Scale (CRBS) questionnaire. It uses a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree), to rate the items. The CRBS includes four subscales: three items about job and time conflicts; five items on logistical issues such as cost, distance, and transportation; nine items concerning perceived needs and healthcare factors; and four related to comorbidities and functional status. Higher ratings indicate more obstacles to enrolling in a CR.
Participation and adherence rate | Day 0, Week 9
  Participation and adherence rates will be documented through self-reflected forms and diaries. Participation rate is defined as the proportion of patients who accepted to participate out of those offered the program, expressed as a percentage. Adherence refers to the proportion of the 24 prescribed trainings attended. Patients attending more than 75% of the total training sessions are considered completers.

CONTACTS AND LOCATIONS:
Overall Officials: Anwar Suhaimi, Principal Investigator — Universiti Malaya Medical Center
Locations (1):
- Universiti Malaya Medical Center, Kuala Lumpur, Lembah Pantai, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 2 months and ending 2 years after the publication of results
Access Criteria: Individual participant data (IPD) underlying published results will be shared with qualified researchers whose analyses aim to advance cardiac rehabilitation science. Requests must include a research proposal detailing objectives, planned analyses, and statistical methods, which may require independent review. Approved applicants must sign a data-sharing agreement. Requests should be submitted to the principal investigator via email. Proposals will be reviewed by a data access committee based on scientific merit, ethical compliance, and consistency with participant consent.